CLINICAL TRIAL: NCT04529083
Title: Feasibility and Functional Outcomes of a Novel Mixed Reality Based System to Manage Phantom Pain for Patients With Lower Limb Amputation.
Brief Title: Mixed Reality Based System to Manage Phantom Pain Phantom Pain for Patients With Lower Limb Amputation
Acronym: MrMAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Collaborators: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Thiru Annaswamy, Staff Physician and Professor, Dallas VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-016
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-03

CONDITIONS: Phantom Limb Pain
Keywords: mixed reality; phantom limb pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Intervention Model Description: Pilot study to evaluate feasibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Mixed Reality System for virtual mirror therapy
  Interventions: Device: Mr. MAPP

INTERVENTIONS:
Device: Mr. MAPP — Mixed reality device to provide virtual mirror therapy to patients with phantom pain

SUMMARY:
The primary goals of this pilot research project are a) to design and develop the a mixed reality based system for managing phantom pain and b) to evaluate the feasibility and preliminary functional outcomes of this system in a sample of patients with lower limb amputation. Findings from this pilot study will serve as preliminary data to inform regarding a fully powered clinical trial to determine the effectiveness and practical implementation of these findings in real-world settings.

Aim1: Design and develop a feasible mixed reality based system to manage phantom pain in patients with lower limb amputation qualifying for on-going mirror therapy.

Hypothesis 1: The investigators hypothesize that the mixed reality based system to manage phantom pain will be feasible and well-received by a sample of patients with lower limb amputation needing mirror therapy.

Aim2: Evaluate functional outcomes in a sample of lower limb amputees (n=10), using this mixed reality based system to manage phantom pain.

Hypothesis 2: Using this system, the investigators hypothesize that patients who participate in the mixed reality based system will show improvements in functional mobility based on performance evaluations and patient reported outcome measures (PROs). The investigators also hypothesize that this mixed reality based system will help to alleviate the phantom pain based on McGill Pain questionnaire and visual analog scale (VAS).

DETAILED DESCRIPTION:
The primary goals of this pilot research project are a) to design and develop the a mixed reality based system for managing phantom pain and b) to evaluate the feasibility and preliminary functional outcomes of this system in a sample of patients with lower limb amputation. Findings from this pilot study will serve as preliminary data to inform regarding a fully powered clinical trial to determine the effectiveness and practical implementation of these findings in real-world settings.

Aim1: Design and develop a feasible mixed reality based system to manage phantom pain in patients with lower limb amputation qualifying for on-going mirror therapy.

Hypothesis 1: The investigators hypothesize that the mixed reality based system to manage phantom pain will be feasible and well received by a sample of patients with lower limb amputation needing mirror therapy.

Aim2: Evaluate functional outcomes in a sample of lower limb amputees (n=10), using this mixed reality based system to manage phantom pain.

Hypothesis 2: Using this system, the investigators hypothesize that patients who participate in the mixed reality based system will show improvements in patient-reported outcome measures (PROs). The investigators also hypothesize that this mixed reality based system will help to alleviate the phantom pain based on Pain questionnaires and visual analog scale (VAS).

Patients 18 years of age and over with history of lower limb amputation and complaint of phantom limb pain. Phantom limb pain is a condition experienced commonly by patients with major limb amputations.

Men and women, over the age of 18 with lower limb amputations (greater than 3 months post surgery) with phantom limb pain.

-Exclusion criteria: ---

* Patients with lower limb amputations with open wounds or active infection in residual or contralateral limbs
* Patients with history of seizures.
* Patients with visual (self-reported) or cognitive impairment (assessed by the mini-mental state examination) that interferes with ability to interact with, participate in, and adhere to a computerized rehabilitation system.
* Any patient with a cardiac event in the last 6 months.
* Any patient with an active medical issue to minimize risk of exacerbating their condition.
* Lives more than 60 miles away from the Dallas VA Medical Center
* Any patient with the motion sickness induced by head mounted displays (HMDs) or immersive environment.
* Any patient experiencing the motion sickness induced by HMDs during the therapy session can also opt out of the study.

In this exploratory, pilot study, a convenience sample of 10 patients will be recruited. A sample of 10 subjects is adequate and consistent with other pilot behavioral intervention trials at the VA that have been completed and published.

This is a pilot study is intended to yield preliminary data that will inform a fully powered trial to determine effectiveness of the novel Mixed Reality based system to manage phantom pain.A HIPAA waiver will be obtained to screen patients with lower limb amputation in the outpatient PM&R clinics. Eligible study candidates will be identified either during an initial visit as an outpatient during clinic visit with the physiatrist. or review of prior visit with physiatrist. The eligible, pre-screened subjects will undergo a basic evaluation (by rehabilitation physician ). After the evaluation, the patient will be asked to participate in the study or sent invitation letter. Once the eligible patient consents to enroll in the study with specific emphasis on safely performing the exercises independently at home. The research team will provide the laptop, camera and instruct the patient in its use at their home. The patient will then use the system and perform the personalized home exercises every day for a 1 month period (to evaluate sustainability of exercise behavior). At the end of this period, the system will be returned. At initial clinic visit, visit at week 1 and 1 month visit, the patient will fill out pain questionnaires, functional questionnaire without any identifiable PHI. The images of the patients performing the exercises will be stored in the encrypted laptop and analyzed at UTD. Also, that the videos at UTD will be destroyed after 5 years, but a copy will be kept at the Dallas VA.

A HIPAA waiver will be obtained to screen patients with lower limb amputation in the outpatient clinics. Eligible study candidates will be identified based on visit as an outpatient, following hospital discharge, the eligible, pre-screened subjects will undergo a basic evaluation (by rehabilitation physician). After the evaluation, the patient will be asked to participate in the study in person or by invitation letter. Once the eligible patient consents to enroll in the study with specific emphasis on safely performing the exercises independently at home. The research team will provide the laptop, camera and instruct the patient in its use at their home. The patient will then use the system and perform the personalized home exercises every day for a 1 month period (to evaluate sustainability of exercise behavior). At the end of this period, the system will be returned by the patient at the final study visit or can be retrieved at subject's home at subjects request if unable to bring to final visit by research assistant. Setting of the Study: The subject will be participating in a therapy session of 15 minutes per day for a duration of 4 weeks. Before starting a session, the subject will be provided with oral instructions about the overall system and the purpose of study. They will be asked to fill out a questionnaire asking the status of phantom pain, phantom limb movement, stress level etc. After completing the questionnaire, they will be allowed to move in virtual world to get acquainted. Each session consists of three sub-sections where the subject is asked to play three different virtual games. These virtual games are designed specifically for lower limb amputees. Each game is targeting certain types of muscle movement. We focused mainly on three types of movements: 1) knee flexion and extension, 2) ankle dorsiflexion and planar flexion, and 3) tandem coordinated bilateral lower extremity movement. Each game will be played only for 5 minutes. After completing each sub-session, the subject is asked to fill out similar questionnaire to record the effect.

System Overview: The system consists of one Microsoft Kinect camera, Oculus Rift and a computer system with sufficient processing power. Microsoft Kinect is used to scan the person and to create corresponding 3D model. As shown in Figure 3, the 3D model for the phantom limb is obtained by mirroring the 3D model of the intact limb. So, the subject will be able to perceive both the limb in the virtual world. The system provides a mixed reality based implementation of mirror therapy for managing phantom pain.

Major features of this system include:

Unconstrained movement: As patient will be performing exercise in virtual environment, the movement is not restricted by limited space as in case of traditional mirror box therapy where user can only move in the limits of box dimension, Realistic illusion of phantom limb: As the Mr.MAPP framework is using RGB-D camera to capture the movement of patients intact limb and mirror it to create the illusion of the phantom limb, the illusion obtained is very realistic instead of using pre-built 3D model of a limb (See Figure 4), Patient Encouragement: Use of an immersive gaming environment motivates and keeps the patient engaging while performing exercise. With the help of virtual reality, various engaging game can be developed that helps to remove monotonousness in therapy sessions.

Feedback with positive Reinforcement: As each game is designed to encourage a patient to perform certain type of exercise, the points earned in the game motivates the patient to perform better, Adherence and compliance monitoring: by recording and annotating the therapy sessions, the coaching software will monitor parameters such as number of repetitions, dates and times of exercises, as well as correctness of performing the exercises. This will serve as a real-time diary which is considered more reliable than self-report diaries that rely on patient recall of activity,Functional Outcome Measures: a) Visual Analog Scale for pain measurement (VAS) and b) McGill Pain questionnaire, c) Additional questions that composite of the Mobility, Activities of Daily Living/Instrumental Activities of Daily Living, and Social Participation.

At the end of the study, the patient will have the option to leave feedback and suggestions for future use of this system.

Descriptive methods will be used to characterize the sample population. Pre-post t-tests or equivalent will be used to compare outcomes at one week and 1 month. Given the pilot nature of this proposed study, inferential statistics (and reporting of statistical significance) will not be used. Feasibility outcomes will be descriptive, including calculating the percent of individuals enrolled in the study versus those eligible and the percent of individuals who remain in the study at month 1. Aims 1 and 2 will help establish intervention acceptability and feasibility. The images of the patients will be stored in the encrypted laptop and analyzed at UTD. Also, that the videos at UTD will be destroyed after 5 years, but a copy will be kept at the Dallas VA .

Using weekly telephone support and online ad-hoc support features of the proposed system, adverse event data will be obtained and further intervention will be initiated as needed for any safety issues that may arise during this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, over the age of 18 with lower limb amputations (greater than 3 months post surgery) with phantom limb pain

Exclusion Criteria:

* Patients with lower limb amputations with open wounds or active infection in residual or contralateral limbs.
* Patients with history of seizures.
* Patients with visual (self-reported) or cognitive impairment (assessed by the mini-mental state examination) that interferes with ability to interact with, participate in, and adhere to a computerized rehabilitation system.
* Any patient with a cardiac event in the last 6 months.
* Any patient with an active medical issue to minimize risk of exacerbating their condition.
* Lives more than 60 miles away from the Dallas VA Medical Center
* Any patient with the motion sickness induced by head mounted displays (HMDs) or immersive environment.
* Any patient experiencing the motion sickness induced by HMDs during the therapy session can also opt out of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gargi Raval, MD, Principal Investigator — North Texas Veterans Healthcare System
Locations (1):
- VA North Texas Health Care System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data may be shared upon approval from concerned authorities if needed

REFERENCES:
- [Derived] Annapureddy D, Annaswamy TM, Raval G, Chung YY, Prabhakaran B. A novel mixed reality system to manage phantom pain in-home: results of a pilot clinical trial. Front Pain Res (Lausanne). 2023 Jun 2;4:1183954. doi: 10.3389/fpain.2023.1183954. eCollection 2023. PMID 37332478
- [Derived] Annaswamy TM, Bahirat K, Raval G, Chung YY, Pham T, Prabhakaran B. Clinical feasibility and preliminary outcomes of a novel mixed reality system to manage phantom pain: a pilot study. Pilot Feasibility Stud. 2022 Oct 22;8(1):232. doi: 10.1186/s40814-022-01187-w. PMID 36273191

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 11
Completed | 8
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: See table below
Arm/Group | Intervention
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Numerical Rating Scale
Description: Pain intensity; 0-10; higher is worse
Time Frame: baseline, 1-month
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 8
score on a scale
  Baseline | 1.75 [1 to 5]
  1-month | 1.125 [1 to 5]
Statistical Analysis 1: Comparison: Intervention; Test type: Other; p = 0.011, t-test, 2 sided; Mean Difference (Net) = -0.625, 95% CI 2-sided [-1.06 to -0.19]

2. Primary Outcome: Change in McGill Pain Questionnaire
Description: Pain intensity and interference; multiple scales; higher is worse. Range 0-78
Time Frame: baseline, 1-month
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 8
score on a scale
  Baseline | 38.5 [0 to 78]
  1-month | 31.88 [0 to 78]

3. Secondary Outcome: Change in Patient Specific Functional Questionnaire
Description: Patient specific functional questionnaire; multiple scales; higher is better; Range 0 to 10 for each activity
Time Frame: baseline, 1-month
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 8
score on a scale
  Baseline | 4.28 [0 to 10]
  1-month | 6.22 [0 to 10]
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p = 0.006, t-test, 2 sided; Mean Difference (Net) = 1.94, 95% CI 2-sided [0.63 to 3.26]

ADVERSE EVENTS:
Time Frame: 1-month
Description: Any difficulties with using the system
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT04529083/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT04529083/ICF_001.pdf